CLINICAL TRIAL: NCT02409186
Title: A Randomized, Controlled, Double-blind Study to Evaluate Efficacy and Survival of Combining Nimotuzumab Plus Concurrent Chemo-radiotherapy in Loco-regional Esophageal Squamous Cell Carcinoma
Brief Title: A Phase III Study of Nimotuzumab Plus Concurrent Chemoradiotherapy in Loco-regional Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NXCEL1311
Record Dates: First submitted 2014-12-03; First posted 2015-04-06 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure | interventions — nimotuzumab; Radiotherapy; Paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab plus chemoradiotherapy (Active Comparator): Nimotuzumab：400mg/w，d1, week 1-7 Paclitaxel：45mg/m2, d1, week 1-7 Cisplatin：20mg/m2, d1, week 1-7 Three dimensional conformal RT（3DCRT）/IntensityModulatedRadiationTherapy（IMRT）：1.8 Gy/f/day, T59.4 Gy/33f,week 1-7
  Interventions: Drug: Nimotuzumab; Radiation: radiotherapy; Drug: chemoradiotherapy Paclitaxel; Drug: chemoradiotherapy Cisplatin
- placebo plus chemoradiotherapy (Placebo Comparator): placebo：400mg/w，d1, week 1-7 Paclitaxel：45 mg/m2, d1, week 1-7 Cisplatin：20 mg/m2, d1, week 1-7 Three dimensional conformal RT（3DCRT）/IntensityModulatedRadiationTherapy（IMRT）：1.8 Gy/f/day, T59.4 Gy/33f,week 1-7
  Interventions: Radiation: radiotherapy; Drug: chemoradiotherapy Paclitaxel; Drug: chemoradiotherapy Cisplatin; Other: placebo

INTERVENTIONS:
Drug: Nimotuzumab — 400mg/w，d1, week 1-7
  Other Names: Taixinsheng
  Arms: Nimotuzumab plus chemoradiotherapy
Radiation: radiotherapy — Three dimensional conformal RT（3DCRT）/IntensityModulatedRadiationTherapy（IMRT）：1.8 Gy/f/day, T59.4 Gy/33f,week 1-7
Drug: chemoradiotherapy Paclitaxel — 45 mg/m2, d1, week 1-7
  Other Names: Paclitaxel
Drug: chemoradiotherapy Cisplatin — 20 mg/m2, d1, week 1-7
  Other Names: Cisplatin
Other: placebo — 400mg/w，d1, week 1-7
  Arms: placebo plus chemoradiotherapy

SUMMARY:
Esophageal cancer is the sixth leading cause of cancer death in worldwide. Over the past 2 decades, well-designed clinical trials have documented the clinical benefits of combination of chemotherapy and radiation for localized esophageal cancer, either as primary therapy or in neoadjuvant setting. Paclitaxel, a radiation sensitizer, has important single-agent activity in esophageal cancer. Paclitaxel-based chemoradiation has been the framework for the recent Radiation Therapy Oncology Group (RTOG) trials of nonoperative management of esophageal cancer. Accumulating clinical evidence suggests that Epidermal Growth Factor Receptor (EGFR) represents a viable target in the treatment of esophageal cancer. EGFR expression is associated with poor prognosis. Nimotuzumab binds specifically to EGFR on both normal and tumor cells and competitively inhibits the binding of Epidermal Growth Factor (EGF) and other ligands, such as Transforming Growth Factor-α (TGF-α). Preclinical models have suggested synergy between nimotuzumab, paclitaxel, cisplatin and radiation. For our phase II study in locally advanced esophageal squamous cell carcinoma (ESCC), the combination of cetuximab and chemoradiotherapy has demonstrated both response and survival benefits. Myara et al reported that nimotuzumab plus concurrent chemoradiation therapy (CCRT) was safe and provided statistically significant objective response (47.8%) and disease control rate (60.9%) in nonresectable ESCC. With all these, the investigators plan to study phase III trial.

DETAILED DESCRIPTION:
The primary endpoint of this study is overall survival, and the primary hypothesis is the experimental arm will improve median survival time (MST) from 18.2 month to 28.5 month. Assuming bilateral ɑ = 0.05, statistical power of 80%.Each group requires a minimum of 59 cases. Consider the 20% loss factor.The total sample size is 200 cases.It is 100 cases in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to study entry
2. age：18-70 years
3. Histopathology confirmed primary esophageal squamous cell carcinoma, meet one of the following criteria (AJCC Staging System，2009，Seventh Edition):Cervical esophageal carcinoma(stage II-III);upper thoracic esophageal cancer or chest esophageal cancer that is unsuitable or refuse surgery (stage II-III)
4. The existence of measurable lesions (according to Response Evaluation Criteria in Solid Tumors 1.1)
5. Eastern Cooperative Oncology Group（ECOG）Performance status of 0-1
6. Possible semi-liquid diet
7. If there is a risk of pregnancy, male and female subjects must be effective contraception during treatment
8. Normal bone marrow reserve: neutrophil (ANC) count≥1500/mm3,platelet count≥100,000 /mm3, hemoglobin≥5.6mmol/L(9g/dL)
9. Normal renal function: serum creatinine≤1.5mg/dl and/or calculated creatinine clearance≥ 60ml/min
10. Normal hepatic function: bilirubin level≤1.5×ULN, alanine aminotransferase aspartate transaminase（ASAT）& ALST≤1.5×ULN
11. Subjects tumor tissue available for the relevant biomarker detection

Exclusion Criteria:

1. Previous chest radiotherapy, systemic chemotherapy, and major esophageal surgery
2. Concurrent chronic systemic immune therapy, targeted therapy, anti-vascular endothelial growth factor（VEGF）therapy or EGFR-pathway targeting therapy not indicated in this study protocol
3. Multiple primary carcinomas of the esophagus
4. Pregnancy (confirmed by urine β-HCG) or lactation period
5. Uncontrolled diabetes, hypertension, and severe cardiac or pulmonary disease
6. There are obvious esophageal ulcers, chest and back more than moderate pain, symptoms of esophageal perforation
7. Unable to comprehend the study requirements or who are not likely to comply with the study requirements
8. Patients with distant metastasis
9. Patients with other malignant disease, except for curable non-melanoma skin cancer, cervical carcinoma in situ or malignant disease cure for≥5 years
10. Known grade 3 or 4 allergic reaction to any of the study treatment
11. Peripheral neuropathy > grade 1
12. Participation in another clinical study within the past 30 days
13. Significant disease which, in the investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Over Survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Ph.D, M.D, Principal Investigator — Shandong Cancer Hospital and Institute; Xue Meng, Ph.D, M.D, Study Director — Shandong Cancer Hospital and Institute
Locations (14):
- China (14):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Guangxi Zhuang Autonomous Region Cancer Hospita, Nanning, Guangxi
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Fourth Hospital of Hebei Medical University Tumor, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Meng X, Zheng A, Wang J, Wu X, Li G, Zhu J, Ma H, Zhu X, Shi A, Dai C, Yan S, Wang B, Qu Z, Han C, Sun X, Ye M, Fan R, Huerxidan N, Wang X, Yu J. Nimotuzumab plus concurrent chemo-radiotherapy in unresectable locally advanced oesophageal squamous cell carcinoma (ESCC): interim analysis from a Phase 3 clinical trial. Br J Cancer. 2023 Nov;129(11):1787-1792. doi: 10.1038/s41416-023-02388-7. Epub 2023 Oct 20. PMID 37864049